CLINICAL TRIAL: NCT01952054
Title: Phase II Study of Denosumab to Define the Role of Bone Related Biomarkers in Breast Cancer Bone Metastasis
Brief Title: Denosumab for Breast Cancer With Bone Mets
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0007; NCI-2014-01273 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-09-20; First posted 2013-09-27 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Breast carcinoma; Bone metastasis; Cancer that has spread to the bone; Denosumab; AMG 162; Prolia; Hormonal agent
MeSH Terms: conditions — Breast Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Denosumab (Experimental): Participants receive a single subcutaneous (SC) administration of Denosumab 120 mg every 4 weeks (+/- 5days). Starting week 5, in addition to receiving Denosumab every 4 weeks, participants receive a hormonal agent chosen by each physician, excluding the agent that participants received at adjuvant therapy setting.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — 120 mg subcutaneously on Day 1 of every 28 day cycle.
  Other Names: AMG 162; Prolia

SUMMARY:
The goal of this clinical research study is to learn if denosumab in combination with a hormonal drug can help lower the number of circulating tumor cells (CTCs) in patients with breast cancer that has spread to the bone. The safety of this combination will also be studied.

This is an investigational study. Denosumab is FDA approved and commercially available to prevent bone-related events caused by breast cancer that has spread to the bone. Using denosumab to lower CTCs in patients with breast cancer that has spread to the bone is investigational.

You may have the option of continuing denosumab after the study ends.

Up to 35 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive denosumab through a needle under your skin on Day 1 of each 28-day study cycle.

Starting on Day 1 of week 4, you will also begin taking a hormonal drug. The study doctor will choose the hormonal drug you receive based on your previous hormonal therapy for breast cancer. The study doctor will give you instructions for taking your hormonal drug.

Study Visits:

On Day 1 of week 4:

* You will have a physical exam
* Blood (about 3 tablespoons) will be drawn for routine tests
* Blood (about 5 teaspoons) will be drawn for CTC testing and to check your immune system.
* Urine will be collected to test for a biomarker that is used to measure the rate of bone breakdown.
* If the study doctor thinks it is needed, you will have a PET scan, a bone scan, or an MRI to check the status of the disease.

On Day 1 of Cycle 2 and Cycle 3, blood (about 1 teaspoon) will be drawn for routine tests.

Length of Study:

You may receive the denosumab and hormonal therapy combination for up to 13 weeks. You will be taken off study if the disease gets worse or intolerable side effects occur.

End of Study Visit:

After your last dose of the study drug, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 3 tablespoons) will be drawn for routine tests.
* Blood (about 5 teaspoons) will be drawn for CTC testing and to check your immune system.
* Urine will be collected to test for a biomarker that is used to measure the rate of bone breakdown.
* If the study doctor thinks it is needed, you will have a PET scan, a bone scan, or an MRI to check the status of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have histological confirmation of breast carcinoma.
2. Patients have progressive metastatic disease with predominantly bone metastasis with 1 or more lesions and at least 1 bone lesion has pathological confirmation, have not been treated or have been treated with any prior therapies (including bisphosphonate treatment and/or radiation therapy). Patients can have soft tissue involvement (Lymph node and skin) and/or metastatic lesions at major organ sites (i.e. lung, liver, etc).
3. Patients have positive ER expression in the primary tumor site by IHC (defined as >/=10%) (PR status is not required)
4. Adequate hematologic function: 1)Absolute neutrophil count (ANC) >/= 1.0 x 10^9/L, 2) Platelet count >/= 50 x 10^9/L, 3) Hemoglobin >/= 9.0 g/dL
5. Adequate cardiac function (LVEF >/= 45%) if patient has known cardiac dysfunction history
6. Adequate Renal function: Calculated creatinine clearance >30 ml/min
7. Adequate Hepatic function: 1) Aspartate aminotransferase (AST) </= 2.5 x ULN; 2) Alanine aminotransferase (ALT) </= 2.5 x ULN; 3) Alkaline phosphatase (Alp) </= 2.5 x ULN; 4) Total bilirubin </= 2.0 x ULN
8. Serum calcium or albumin-adjusted serum calcium >/=2.0mmol/L (8.0mg/dL) and </= 2.9 mmol/L (11.5mg/dL)
9. Patients have ability and willingness to sign written informed consent.
10. Patients are 18 years of age or older.
11. Female patients of childbearing potential (A female not free from menses > 2 years or not surgically sterilized) must be willing to use highly effective contraception to prevent pregnancy or agree to abstain from heterosexual activity throughout the study. Highly effective contraception, defined as male condom with spermicide, diaphragm with spermicide, intra-uterine device. Highly effective contraception must be used by both sexes during the study and must be continued for 5 months after the last dose of denosumab.
12. Female patients of childbearing potential must have negative serum pregnancy test </= 21 days prior to starting study treatment.
13. Patients have CTC >/=3.

Exclusion Criteria:

1. Patients have known sensitivity to any of the products to be administered during the study (e.g., mammalian derived products, calcium, or vitamin D).
2. Patients receiving concurrent anti-cancer therapy (chemotherapy, immunotherapy, radiation therapy and biological therapy) while taking study medication. However, patients receiving CDK4/6 inhibitor or mTOR inhibitor as a standard of care while on study is permitted.
3. Patients with metastatic sites that requires chemotherapy.
4. Patients with active infection and requiring IV or oral antibiotics.
5. Patients with concurrent disease or condition that would make them inappropriate for study participation, or any serious medical disorder that would interfere with patients' safety.
6. Patients have HER2-positive breast carcinoma (IHC staining more than 3+ or HER2 gene amplification by FISH)
7. Patient is pregnant or breast feeding, or planning to become pregnant within 5 months after the end of treatment.
8. Patient is of child bearing potential and is not willing to use, in combination with her partner, two highly effective methods of contraception or abstinence during treatment and for 5 months after the end of treatment.
9. Male patients.
10. Patients have prior history or current evidence of osteonecrosis/osteomyelitis of the jaw.
11. Patients have active dental or jaw condition which requires oral surgery, including tooth extraction.
12. Patients have non healed dental/oral surgery, including tooth extraction.
13. Patients planned invasive dental procedures.
14. Patients experiencing a visceral crisis including severe organ dysfunction as assessed by > Gr 2 symptomatic toxicities, laboratory studies, and/ or rapid progression of disease originating from visceral metastasis.
15. Patients that have received the study medication (Xgeva/Prolia).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 8, 2015 to Apr 4, 2017. All recruitment performed at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: One participant was ineligible due to screen failure
Groups:
- Denosumab: Subcutaneous administration of Denosumab 120 mg every 4 weeks (+/- 5days). Starting week 5, also receive a hormonal agent chosen by physician.
Period: Overall Study
Arm/Group | Denosumab
Started | 6
Completed | 5
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Denosumab
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Denosumab in Reducing Circulating Tumor Cells (CTCs) Among Breast Cancer Patients With Bone Metastases.
Description: The difference in number of CTCs in 7.5 ml whole blood from baseline to week4. CTC reduction from baseline to week4 is statistically analyzed using the two-sided paired t-test with the significance level of 0.05.
Time Frame: Baseline, week 4
Population: The primary objective could not be met due to technical issues.
Arm/Group | Denosumab
Number analyzed (Participants) | 0

2. Secondary Outcome: The Changes of Epithelial-mesenchymal Transition (EMT) in CTCs
Description: The change in Her2, Muc-1, GA733-2 (EpCAM), Twist, Akt, PI3K and ALDH-1 in CTCs after 1 st cycle of treatment with denosumab.
Time Frame: Baseline, week 4
Measure: Mean (Standard Deviation); unit: ng/uL
Arm/Group | Denosumab
Number analyzed (Participants) | 6
ng/uL
  HER 2 | .003 (.032)
  Muc-1 | .065 (.062)
  GA733-2 (EpCAM) | -.372 (.750)
  Twist | .018 (.045)
  Akt | .028 (.077)
  ALDH-1 | .328 (.808)

3. Secondary Outcome: The Changes in Urine N-telopeptide Level
Description: The collection urine is performed at baseline, at week4 and the end of 3rd cycle (week13) to evaluate the level of N-telopeptide.
Time Frame: Baseline up to week 13
Measure: Mean (Standard Deviation); unit: nmol/mmol
Arm/Group | Denosumab
Number analyzed (Participants) | 6
nmol/mmol
  Baseline | 59.0 (59.0)
  Week 4 | 19.3 (7.7)
  Week 13 | 21 (9.5)

ADVERSE EVENTS:
Time Frame: Through study completion 13 weeks
Description: A serious adverse event is any adverse drug experience occurring at any dose that results in any of the following outcomes: Death, a life-threatening adverse drug experience, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity and a congenital anomaly/birth detect. One participant was ineligible due to screen failure.
Arm/Group | Denosumab
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab (N=6)
Constipation (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neutrophil count decreased (Investigations) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Fatigue (General disorders) | 2
Anxiety (Psychiatric disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Headache (Nervous system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Agitation (Psychiatric disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Bladder infection (Infections and infestations) | 1
Dizziness (Nervous system disorders) | 1
Edema limbs (General disorders) | 1
Eye disorders-other specify-red/burning, tearing eyes (Eye disorders) | 1
Eyelid function disorder (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fever (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Hot Flashes (Vascular disorders) | 1
Insomnia (Psychiatric disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT01952054/Prot_SAP_000.pdf